CLINICAL TRIAL: NCT02992951
Title: A Randomised Controlled Trial to Assess the Clinical and Cost Effectiveness of Dialkylcarbamoylchloride (DACC) Coated Post-operative Dressings Versus Standard Care in the Prevention of Surgical Site Infection in Clean or Clean-contaminated, Vascular Surgery.
Brief Title: DACC in the REduction of Surgical Site INfection
Acronym: DRESSINg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R2034
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2026-01-30 (Actual); Status verified 2025-05

CONDITIONS: Infection, Bacterial; Wound Infection; Wound Infection, Surgical; Surgical Incision; Surgical Wound
Keywords: Infection; Surgical Site Infection; Dialkylcarbamoylchloride
MeSH Terms: conditions — Bacterial Infections; Wound Infection; Surgical Wound Infection; Surgical Wound; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DACC-Coated Post-Operative Dressing (Experimental): DACC-Coated Post-Operative Dressing
  Interventions: Device: DACC-Coated Post Operative Dressing
- Non-DACC coated Occlusive Post-operative Film Dressing (No Intervention): Non-DACC coated Occlusive Post-operative Film Dressing

INTERVENTIONS:
Device: DACC-Coated Post Operative Dressing — Leukomed Sorbact is a non-active coated wound dressing, containing Dialkylcarbomoylchloride. This is a bacteria-binding compound that adheres bacteria via hydrophobic interaction and removes them from the wound bed at dressing change.
  Other Names: Leukomed Sorbact
  Arms: DACC-Coated Post-Operative Dressing

SUMMARY:
Surgical site infection is an infection at a place in the body where surgery has taken place, and has been reported in around 5% of people undergoing an operation. In vascular surgery, infection rates are as high as 30%. Methods to reduce this rate of infection should be investigated thoroughly for their effectiveness and cost-effectiveness.

The investigators aim to conduct a research trial examining one such method. Leukomed Sorbact is a wound dressing coated with a chemical (DACC) derived from spider-silk that interacts with, and binds bacteria, causing them to be mechanically removed from a wound when the dressing is changed. The trial aims to compare the effectiveness of this dressing to a standard, non-coated dressing, in the reduction of surgical site infection.

718 patients from a number of centres across the UK will be recruited to this study. Adult patients who are having a vascular surgery operation will be approached for entry into the trial. The trial will be explained to them, as well as an explanation that participation is voluntary and their operation or other aspects of their care will not be impacted in any way should participants not wish to participate.

Participants will be randomised by computer into one of two groups - one group whose wounds are dressed with Leukomed Sorbact, and the other whose wounds are dressed with a standard dressing. Patients will be followed up at 30 days post-operatively. At the follow up, their wounds will be inspected for infection, and participants will be asked to complete short questionnaires measuring quality of life. Quality of life will also be assessed at 3 months post surgery.

The trial will aim to answer a number of questions, with the primary question being does a DACC coated dressing applied after an operation reduce the risk of an infection at the surgery site? It will also ask whether this treatment is cost-effective and whether it promotes satisfactory healing and evaluate the overall carbon footprint impact of each intervention.

Studies Within a Trial will be conducted to validate a remote diagnostic measure for detecting surgical site infection using wound images and the Bluebelle Wound Healing Questionnaire, evaluate feasibility of novel hair removal methods such as epilation and waxing, carbon footprint modelling within randomised controlled trials.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for inclusion in the study the participants must meet the following criteria:

* Adults ≥18 yrs undergoing clean or clean-contaminated lower limb vascular surgery, with wounds closed by primary intention.
* Able to understand the Patient Information Sheet and supplementary materials and capable and willing to give informed consent and follow the protocol requirements (including attending all follow-up visits and completing written questionnaires).

Exclusion Criteria:

Patients will not be included in the study if they meet any of the following exclusion criteria:

* Patients on antibiotics for other conditions at the time of surgery or in the follow up period.
* Patients undergoing any procedure that does not include lower limb incisions.
* Allergies to any component of either the DACC-coated dressing or the control dressing.
* Inability to give informed consent due to incapacity (as defined by the MCA 2005)
* Aged under 18 years at the time of recruitment
* Use of investigational drug/device therapy within preceding 4 weeks that may interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2025-06-28 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
30 day infection rate | 30 days
  Surgical Site Infection at 30 days post-op

SECONDARY OUTCOMES:
3 month infection rate | 3 months
  Surgical Site Infection at 3 months post-op (implant patients only)
Quality of Life (SF-36 V2) | 30 days, 3 months
  Score ranging from 0-100, higher values indicating better health
Quality of Life (EQ-5D-3L) | 30 days, 3 months
  Score ranging from 5-15, higher scores indicating worse health
Mortality | 30 days
  30-day mortality
Bluebelle wound healing questionnaire | Days 30 and 37
  Score ranging 0-41, higher values indicating infection
Carbon Footprint Analysis | 3 months
  Healthcare resource use data

OTHER OUTCOMES:
SWAT 1 Validation Acceptability | 30 and 37 days
  Response rates to measure at 30 and 37 days
SWAT 1 Validation reliability | 30 and 37 days
  Inter and intra rater reliability
SWAT 1 Validation Validity | 30 days
  Sensitivity, specificity, ROC analysis, AUC
SWAT 2 Hair Removal Feasibility | 30 days
  Safety/adverse events
Carbon Footprint Model Development | 3 months
  Healthcare resource use data, consumable item weights

CONTACTS AND LOCATIONS:
Overall Officials: George Smith, M.D, Principal Investigator — Hull University Teaching Hospitals NHS Trust
Locations (1):
- Academic Vascular Surgery Unit, Vascular Laboratory, Alderson House, Hull Royal Infirmary, Hull, East Riding of Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Totty JP, Harwood AE, Cai PL, Hitchman LH, Smith GE, Chetter IC. Assessing the effectiveness of dialkylcarbamoylchloride (DACC)-coated post-operative dressings versus standard care in the prevention of surgical site infection in clean or clean-contaminated, vascular surgery (the DRESSINg trial): study protocol for a pilot feasibility randomised controlled trial. Pilot Feasibility Stud. 2019 Jan 18;5:11. doi: 10.1186/s40814-019-0400-2. eCollection 2019. PMID 30680225
- [Derived] Cristino MA, Nakano LC, Vasconcelos V, Correia RM, Flumignan RL. Prevention of infection in aortic or aortoiliac peripheral arterial reconstruction. Cochrane Database Syst Rev. 2025 Apr 22;4(4):CD015192. doi: 10.1002/14651858.CD015192.pub2. PMID 40260835
- See also: Abstract Link — https://pilotfeasibilitystudies.biomedcentral.com/articles/10.1186/s40814-019-0400-2